CLINICAL TRIAL: NCT04151953
Title: Evaluation of Potential Myocardial Injury in Patients With Cardiac Implantable Electronic Devices Following Magnetic Resonance Imaging
Brief Title: Myocardial Injury in Patients With Cardiac Implantable Electronic Devices Following Magnetic Resonance Imaging
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Allan S. Jaffe, Principal Investigator, Mayo Clinic
Other Study IDs: 19-004286
Record Dates: First submitted 2019-11-02; First posted 2019-11-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Magnetic Resonance Imaging (MRI)
Keywords: Pacemaker; Implantable Cardioverter Defibrillator (ICD); Cardiac implantable electronic device (CIED)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum or plasma samples remaining after initial analysis will be frozen and stored at -80 degrees Celsius for 120 months (10 years). These samples may be used if there are new and more sensitive biomarkers of myocardial injury that become available.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with cardiac implantable electronic device (CIED): Subjects with previously implanted cardiac implantable electronic device (CIED) who are undergoing an MRI Scan for clinically indicated, diagnostic purposes.
  Interventions: Diagnostic Test: Blood sample collection

INTERVENTIONS:
Diagnostic Test: Blood sample collection — Blood sample collection for markers of myocardial injury

SUMMARY:
Researchers are trying to determine if heart injury occurs in subjects with cardiac implantable electronic device (CIED), such as a pacemaker or implantable cardioverter defibrillator (ICD), who undergo a magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
With an aging population and growing indications for both MRI and CIEDs, it is estimated that patients with a CIED will have up to a 75% likelihood to meet some indication for MRI during their lifetime. MRI in patients with CIEDs has been increasingly shown to be a viable option in a variety of clinical circumstances under strict protocols and close monitoring. It is uncertain if MRI results in myocardial injury. Injury could occur due to heating of the lead(s) with myocardial heating and injury occurring at the lead tip.

A previous Mayo study published in 2016 showed no significant changes in cardiac troponin levels in the majority of patients with a CIED when MRI was performed. This study however was done using the older, less sensitive troponin assay. Unpublished data from the Mayo ED showed an increase in diagnosis of acute myocardial injury from 39% to 62% after implementation of the new hs-cTnT assay, reflecting its increased sensitivity. The previous Mayo study was also a retrospective study, and thus the data gathered was not as rigorously controlled as might be ideal.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have CIED devices (whether conditional or unconditional, regardless of the type of device e.g. ICD, pacemakers, leadless pacemakers) who undergo MRI for any reason

Exclusion Criteria:

* Patients under age 18
* Patients with myocardial infarction, coronary artery bypass grafting or any invasive cardiac procedure in the previous six weeks
* Pregnant patients
* Patients who cannot provide informed consent because of cognitive dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult males and females age 18 and above identified from the electronic medical record (EMR) calendar of patients with devices who are coming for a MRI
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Myocardial injury | Baseline, 6-24 hours post MRI
  Changes in high sensitivity cardiac troponin T (hs-cTnT) or troponin I (hs-cTnI) assay

CONTACTS AND LOCATIONS:
Overall Officials: Allan S Jaffe, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials